CLINICAL TRIAL: NCT05381506
Title: A Phase II, Prospective, Multicenter Study Ofrelabrutinib in Combination With Gemox in Refractory / Relapsed Diffuse Large B-cell Lymphoma
Brief Title: Study of Orelabrutinib in Combination With Gemox in Refractory / Relapsed Diffuse Large B-cell Lymphoma
Acronym: O-Gemox
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhiming, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-FXY-102-内科
Record Dates: First submitted 2022-05-15; First posted 2022-05-19 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-05

CONDITIONS: DLBCL
Keywords: Orelabrutinib; Gemox
MeSH Terms: interventions — orelabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Orelabrutinib and Gemox (Experimental): Orelabrutinib and Gemox for 6 cycles
  Interventions: Drug: Orelabrutinib and Gemox

INTERVENTIONS:
Drug: Orelabrutinib and Gemox — Drug: Orelabrutinib Orelabrutinib 200mg, po, qd
  Drug: Gemox14 Gemcitabine, Oxaliplatin
  Other Names: O-Gemox

SUMMARY:
This study aims to investigate the treatment of refractory or relapsed DLBCL with orelabrutinib and gemox. The primary endpoint is response rate (complete response rate and overall response rate), and the second endpoints are survival time (OS and PFS) and toxicities.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed relapsed or refractory Diffuse Large B-cell Lymphoma. There must be at least one evaluate able or measurable lesion that meets the Lugano criteria
2. Age beyond18 years old;
3. ECOG performance status 0-2.
4. Estimated survival time > 12 weeks.
5. Adequate first-line treatment with CD20-containing monoclonal antibody
6. DLBCL patients confirmed as non-GCB by Han's classification
7. The main organs function well, namely, the following requirements were met one week before admission: Blood routine ANC ≥ 1.5×109/L, Hb ≥ 100g/L and PLT ≥ 100×109/L; liver function were normal (total bilirubin ≤1.5×ULN, ALT and AST ≤ 2.5×ULN), renal function was normal (serum creatinine ≤1×upper limitation of normal (ULN)), and without abnormal coagulation function.
8. Pregnant women of childbearing age must have a pregnancy test (serum or urine) within 14 days before enrollment and the result is negative, and they are willing to use reliable methods of contraception during the test.
9. The subjects who volunteer to join the study and sign the informed consent form, have good compliance and cooperate with the follow-up.

Exclusion Criteria:

1. Patients with central nervous system involvement
2. Patients with Myc gene and BCL2/BCL6 gene rearrangement at the same time;
3. Patients who have received BTK inhibitor therapy in the past;
4. Patients who have received Gemox or GDP chemotherapy in the past;
5. History of other malignancy within the last 5 years prior to enrollment, except for cured basal cell carcinoma of skin, cervix in situ carcinoma and superficial bladder cancer;
6. Suffering from the following cardiovascular diseases: myocardial ischemia or myocardial infarction above grade II, poorly controlled arrhythmia (including QTc interval ≥ 450 ms for men and ≥ 470 ms for women); according to NYHA standards, grades III to IV cardiac function Incomplete, or echocardiography showed left ventricular ejection fraction (LVEF) <50%;
7. Abnormal coagulation function (INR>1.5 or prothrombin time (PT)>ULN+4 seconds or APTT>1.5 ULN), with bleeding tendency or receiving thrombolysis or anticoagulation therapy;
8. Arterial/venous thrombotic events, such as cerebrovascular accident (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep venous thrombosis and pulmonary embolism, that occurred within 12 months before enrollment;
9. Known hereditary or acquired bleeding and thrombotic tendencies (such as hemophiliacs, coagulation disorders, thrombocytopenia, hypersplenism, etc.);
10. Received major surgical operation or suffered severe traumatic injury, fracture or ulcer within 4 weeks of enrollment;
11. There are factors that obviously affect the absorption of oral drugs, such as inability to swallow, chronic diarrhea and intestinal obstruction;
12. Active infection requires antimicrobial treatment (for example, antibiotics and antiviral drugs are required, excluding chronic hepatitis B, anti-hepatitis B treatment, and antifungal drug treatment);
13. Active hepatitis B (HBV DNA ≥ 2000IU/mL or 104 copies/mL) or hepatitis C (positive hepatitis C antibody, and HCV RNA is higher than the detection limit of the analytical method);
14. Those who have a history of psychotropic substance abuse and cannot quit or have mental disorders;
15. Participated in clinical trials of other anti-tumor drugs within 4 weeks before enrollment;
16. Received strong CYP3A4 inhibitor treatment within 7 days before enrollment, or received strong CYP3A4 inducer treatment within 12 days before participating in the study;
17. Pregnant or breastfeeding women; fertile patients who are unwilling or unable to take effective contraceptive measures;
18. The investigator judges other circumstances that may affect the conduct of clinical research and the judgment of research results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 12 weeks after the initiation of the treatment
  overall response rate after treated by Orelabrutin and Gemox

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to two years after the start of the study
  PFS was defined as time from study registration to first disease progression or death whichever occurred first, otherwise subject data were censored at time last known disease free
Overall Survival (OS) | Up to two years after the start of the study
  OS was defined as time from study registration to death, and otherwise censored at time last known alive
Duration of Response（DOR） | Up to three years after the start of the study
  The time from the first assessment of CR or PR to PD (progressive disease) or death from any cause
Adverse events | Up to one year after the start of the study
  All the adverse events of the patients related will be assessed and graded by NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Zhiming Li, Dr., Study Chair — Sun Yat-sen University
Locations (8):
- China (8):
  - Chongqing Cancer Hospital, Chongqing, Chongqing Municipality
  - Guangxi Medical University Cancer Hospital, Naning, Guangxi
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - West China Hospital.Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang